CLINICAL TRIAL: NCT02186665
Title: A Multicenter, Randomized, Double Blind, Parallel Group, Vehicle Controlled, Study of the Safety and Efficacy of Calcitriol 3 mcg/g Ointment Applied Twice Daily for 8 Weeks in Pediatric Subjects (2 to 12 Years of Age) With Mild to Moderate Plaque Psoriasis
Brief Title: Plaque Psoriasis Study in Pediatric Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18132
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2017-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- calcitriol ointment (Experimental): calcitriol 3 mcg/g ointment
  Interventions: Drug: calcitriol ointment
- placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: calcitriol ointment
  Arms: calcitriol ointment
Drug: placebo comparator
  Arms: placebo

SUMMARY:
The purpose of this study is to compare the safety, efficacy and calcium metabolism of up to 8 weeks of treatment with calcitriol 3 mcg/g ointment versus its vehicle, when used twice daily, without occlusion, to treat children aged 2 to 12 years, with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 2 to 12 years of age
* Clinical diagnosis of stable mild to moderate plaque psoriasis

Exclusion Criteria:

* Other forms of psoriasis
* Hypercalcemia
* Past history of kidney stones
* Vitamin D deficiency
* Other concomitant dermatological disease

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D, LLC
Locations (34):
- United States (12):
  - David Stoll, MD, Beverly Hills, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Dermatology Specialists Research, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - RCMC Center for Dermatology at Linden Oaks, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - DermResearch, Austin, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Jordan Valley Dermatology, West Jordan, Utah
- Belgium (3):
  - UCL Saint Luc, Brussels
  - UZ Ghent, Ghent
  - CHU de Liège, Liège
- Winnipeg Clinic, Dermatology Research, Winnipeg, Manitoba, Canada
- Germany (5):
  - Universitätsklinikum Erlangen, Hautklinik, Erlangen
  - Praxis Dr.Beate Schwarz, Langenau
  - Universitäts-Hautklinik Mainz, Johannes Gutenberg-Universität Mainz, Mainz
  - Technical University Munich, München
  - University of Tübingen, Tübingen
- Hungary (3):
  - Heim Pál Gyermekkórház; Bőrgyógyászati Osztály, Budapest
  - Pécsi Tudományegyetem; Bőr-, Nemikórtani és Onkodermatológiai Klinika, Pécs
  - Szegedi Tudományegyetem, Szent-Györgyi Albert Klinikai Központ; Bőrgyógyászati és Allergológiai Klinika, Szeged
- Italy (4):
  - PO G. Rodolico, AOU Policlinico Vittorio Emanuele, Catania
  - Padova University Hospital, Padua
  - University of Parma, Parma
  - Policlinico Tor Vergata, Rome
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona-Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcitriol Ointment | Placebo
Started | 8 | 11
Completed | 8 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcitriol Ointment | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.8) | 9.8 (1.8) | 9.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Success of Investigator's Global Assessment (IGA)
Description: The number of subjects with a minimum improvement of 2 grades from baseline in the IGA score and a severity rating of 0 (clear) of 1 (almost clear) at Week 8 (LOCF).
  The IGA was evaluated at each visit on the following 0 to 4 point scale:
  0 - Clear: No signs of psoriasis except for residual hypopigmentation / hyperpigmentation
  1. - Almost Clear: Just perceptible erythema, no induration, and no scaling
  2. - Mild: Mild erythema, no induration, and mild or no scaling
  3. - Moderate: Moderate erythema, mild induration, and mild or no scaling
  4. - Severe: Severe erythema, moderate to severe induration, and scaling of any degree
Time Frame: Baseline to Week 8
Population: ITT: All randomized subjects to whom study medication was dispensed.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcitriol Ointment | Placebo
Number analyzed (Participants) | 8 | 11
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Calcitriol Ointment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 6/8 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol Ointment (N=8) | Placebo (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Conjuctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lice infestation (Infections and infestations) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (2)
Urine calcium/creatinine ratio increased (Investigations) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No